CLINICAL TRIAL: NCT06972979
Title: A Randomized Trial of Gamification and Remote Support to Improve Statin Adherence
Brief Title: Investigation of a Patient Support Intervention for Statin Medication Adherence
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ascension Health (Industry)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mitesh Patel, Chief Clinical Transformation Officer, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: RAS20250009
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Medication Adherence
Keywords: Gamification; Remote Support; Statin; Adherence; Primary Care
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized, controlled trial to test the effectiveness of a behaviorally-designed gamification intervention with remote nursing support to increase statin adherence after 6-months. Patients will be randomized after they opt-in and consent for the program within the following Ascension states: FL, IN, TN, TX.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Participants in the usual care arm will have consented for participation and will be informed they are on a waiting list for approximately 6-12 months. During that time they will receive no additional interventions beyond usual care and not be be invited again to enroll in the MedTrack program.
- Text Message Group (Experimental): Participants in the intervention arm will have consented for participation in the MedTrack program and will receive the text message intervention and remote support within 1-2 weeks of enrolling.
  Interventions: Behavioral: Text Message Gamification and Remote Support

INTERVENTIONS:
Behavioral: Text Message Gamification and Remote Support — Participants in the intervention arm consists of several components: (I) medication check-ins with the ability to set the time(s) for daily medication reminders, (II) a gamification experience to drive behavior change, (III) ability to identify a support partner who receives weekly updates on the patient's game status; (IV) access to an RN team for clinical questions and care coordination, and (V) patients' providers can see real-time progress within an electronic health record (EHR) integrated application.
  Arms: Text Message Group

SUMMARY:
Statins have been demonstrated to significantly reduce the risk of cardiovascular disease, but adherence to these medications is suboptimal. Improving adherence can be challenging because it is multifactorial and behaviors often occur within the everyday lives of patients and are less addressable during a visit with a clinician. In this study, the investigators will conduct a randomized trial to evaluate a behaviorally-designed gamification intervention with remote nursing support to improve statin adherence.

DETAILED DESCRIPTION:
Improving medication adherence can be challenging because behaviors occur within the everyday lives of patients. Therefore, intermittent visit-based adherence interventions or refill reminders have had limited impact. Remote Patient Monitoring (RPM) has been demonstrated in other settings to improve daily health behaviors when combined with automated outreach and a behavioral change strategy, such as gamification. These approaches have been demonstrated to be effective for other daily behaviors such as increasing physical activity levels among a wide range of patient populations including those at elevated risk for major cardiovascular events. MedTrack is a text message-based remote patient monitoring program with several key components: (I) medication check-ins with the ability to set the time(s) for daily medication reminders, (II) a gamification experience to drive behavior change, (III) ability to identify a support partner who receives weekly updates on the patient's game status; (IV) access to an RN team for clinical questions and care coordination, and (V) patients' providers can see real-time progress within an electronic health record (EHR) integrated application.

ELIGIBILITY:
Inclusion Criteria:

* Adults, age 18 and older
* Have a mobile phone number or email on file to receive a digital outreach to participate in the study
* Have a primary care provider (PCP) employed by Ascension.
* Prescribed a statin medication and had filled two statin prescriptions in the previous 12 months (one in the prior 6 months and another in the previous 6 to 12 months)
* PDC <80% in the prior 12 months
* Have consented for electronic communications with Ascension

Exclusion Criteria:

* Patients will be excluded if they do not meet our inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2200 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Statin adherence, population average | 6-months after enrollment
  Statin adherence, measured using the proportion of days covered (PDC), during the 6-month intervention period

SECONDARY OUTCOMES:
Statin adherence, proportion of population with PDC>=80% | 6-months after enrollment
  Proportion of patients with statin PDC adherence greater than or equal to 80% during the 6-month intervention period

CONTACTS AND LOCATIONS:
Locations (1):
- Ascension Health, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The study has patient information that the investigators are not approved to share.